CLINICAL TRIAL: NCT06499064
Title: Information and Communications Technology (ICT)-based Modeling of Transthyretin-associated Amyloidosis Cardiomyopathies (ATTR-CM) Care: EOSS-ATTR Study (eHealth Based Operative Support System in ATTR-CM)
Brief Title: EOSS-ATTR Study (eHealth Based Operative Support System in ATTR-CM)
Acronym: eOSS-ATTR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Sergi Yun, Internal Medicine Specialist. MD. Principal investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IDIBELL-PR361/23
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Amyloid Cardiomyopathy; ATTR Amyloidosis Wild Type; ATTR Gene Mutation
Keywords: eHealth; mHealth; telemonitoring; ATTR, heart failure
MeSH Terms: conditions — Heart Failure; Amyloid Neuropathies, Familial | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth (Experimental): Structured follow-up in the basis of using mHealth-based solution. mHealth will include daily signs and symptoms telemonitoring and structured follow-up by the means of video or audio-conference.
  Interventions: Procedure: mHealth
- Usual care (No Intervention): Patients with usual care follow-up in a heart failure due to ATTR-CM program.

INTERVENTIONS:
Procedure: mHealth — Follow-up and treatment of patients in the mHealth arm will be based on a comprehensive solution for the care and monitoring of chronic patients, modelled and tested in chronic HF patients. This is the PIRENe platform, previously described and evaluated in HF patients. It is a digital solution, external to the centre's information systems (external platform). However, it has some special features in its design in terms of remote monitoring, educational tools, among others, expressly conceived and designed for patients with ATTR-CM. This platform allows the provision of multichannel service and monitoring of patients through:
  1. Patient monitoring of: Biometric data and symptom report.
  2. Generation and management of warning alarms notified to the professionals assigned to each patient in case one of the following situations occurs.
  3. Follow-up via videoconference.
  Arms: mHealth

SUMMARY:
Unicenter, proof-of-concept, prospective, randomised, controlled, open-label and blinded end-point adjudication trial to assess the effect on patient-reported outcomes measures (PROMs), patient-reported experience measures (PREMs) and clinical events of a mHealth-based comprehensive management program for patients with chronic heart failure (HF) due to transthyretin-associated amyloidosis (ATTR)-cardiomyopathy (CM) by means of remote daily telemonitoring of signs and symptoms and remote structured follow-up using videoconference.

DETAILED DESCRIPTION:
Background and Rationale:

Early diagnosis as well as optimal care of transthyretin-associated amyloidosis (ATTR)-cardiomyopathy (CM) is crucial to improve the outcome of these patients. In order to perform a personalised and patient-centred ATTR-CM, it is essential to integrate new advanced diagnostic and monitoring tools to the pre-existing ones. In this regard, electronic health (eHealth)-based solutions have been gradually being incorporated into the follow-up of chronic patients (e.g. heart failure [HF] patients, among others) over the last few years.

Objectives:

The main objective of this study is to improve the process of care, diagnosis and monitoring of the patient with ATTR-CM by means of a multidisciplinary and transversal model using new digital technologies and optimizing work processes (eHealth-based healthcare management). The primary objective of the study will be the changes in patient-reported outcomes (PROMs) such as self-care and quality of life (QoL) between patients followed and monitored using the mHealth-based digital tool (mHealth) and those in standard follow-up (usual care [UC]). Key secondary objectives will include changes in patient-reported experience measures (PREMs), the occurrence of events, among others between those with and without mHealth-base-ATTR management.

Methodology:

The eOSS-ATTR study will be a study with 2 phases: i) #Phase 1: a design, implantation and pre-clinical evaluation of the digital platform; and ii) #Phase 2: a subsequent clinical evaluation phase. The clinical phase (#Phase 2) will be a unicenter, proof-of-concept, prospective, randomised, controlled, open-label and blinded end-point adjudication trial to assess the effect on PROMs, PREMs and clinical events of a mHealth-based comprehensive management program for patients with HF due to ATTR-CM by means of remote daily telemonitoring of signs and symptoms and remote structured follow-up using videoconference. Regarding #Phase 1, it is proposed to evolve the MAST (Model for Assessment of Telemedicine) model, adding the consideration of the stakeholders involved in the use of this technology, as well as the different use cases and scenarios. All assessed items will be compared before and after the eHealth solution implementation. Concering #Pase 2, HF patients due to ATTR-CM with a HF decompensation in the last 12 months will be randomised (1:1) to structured follow-up based on face-to-face appointments (UC group) or the delivery of health care using mHealth (mHealth group). Randomisation will be stratified at each ATTR subtype (variant [ATTRv] or wild-type form [ATTRwt] and according to the presence or absence of frailty to ensure balanced assignment of frail patients to each group. The follow-up will be of 6 months in two groups and will be nurse-led and based on mHealth solution designed and modeled for the follow-up of patients with ATTR-CM in the mHealth group. This technological solution is proposed to improve the care monitoring and outcomes of ATTR-CM patients. Patients will be recruited for 12 months.

Expected Results:

eOSS-ATTR study is the first trial to integrate and assess mHealth solutions combining telemonitoring and structured teleintervention via videoconference in 'real-world' HF patients due to ATTR-CM to improve clinical outcomes and new clinical events. Its great value is that it assesses 'real-world' patients in terms of frailty, comorbidity, literacy level, skills with new technologies among others. Such strategies are of enormous value for the prognosis, QoL and experience of patients with HF due to ATTR-CM. Integration of solutions based on mHealth into day-to-day HF monitoring with user-friendly technology that provides the possibility of direct contact with their care team can contribute to a clear clear improvement in PROMs and PREMs as well as a reduction of new clinical events. It will allow us to optimise the care of HF due to ATTR-CM patients in this period in terms of self-care education as well as treatment optimisation and empowerment in disease management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* HF diagnosis according to European Society of Cardiology (ESC)
* Patients with a HF decompensation in the last 12 months
* Confirmed diagnosis of ATTR-CM (ATTRv or ATTRwt)
* Written informed consent

Exclusion Criteria:

* Age<18 years old
* Participation in another clinical trial
* Moderate or severe cognitive impairment without a competent caregiver
* Lack of social support
* Institutionalized patients
* Life expectancy less than 1 year (excluding HF)
* Institutional-based or end-of-life care
* Serious psychiatric illness
* Planned cardiac surgery
* Planned heart transplantation or left ventricular assist device (LVAD) implant
* Patients in haemodialysis program
* The patient is unable or unwilling to give the informed consent to participate
* The patient is considered an unsuitable candidate for this study according to the decision of the local investigator
* Unstable patients with signs of fluid overload or low cardiac output

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of self-care using a validated scale (European Heart Failure Self-Care Behavior Scale). | Six months after inclusion of the patient
  changes in patient-reported outcomes (PROMs) such as self-care European Heart Failure Self-Care Behaviour Scale) between patients followed and monitored using the mHealth-based digital tool (mHealth) and those in standard follow-up (usual care [UC]).
Improvement of quality of life using a validated questionnaire (EUROQOL - 5D). | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.

SECONDARY OUTCOMES:
Occurrence of new clinical events (readmission [all-cause, HF, CV and non-CV] rate and total number; worsening HF events; urgent HF visits; all-cause, CV and non-CV death). | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Incidence of implantation of devices (pacemakers, cardiac resynchronization therapy [CRT] or implantable cardioverter defibrillator [ICD]) | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Change of NYHA functional class | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Change of 6-minutes walking test [6MWT] distance. | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Evolution of ATTR-CM stages | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Changes in prognostic biomarkers: atrial natriuretic peptide levels (brain natriuretic peptide [BNP] and/or N-terminal-pro-brain natriuretic peptide [NT-proBNP]) and troponin levels (troponin T [TnT] and/or troponin I [TnI]). | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.
Improvement of patient reported experience measures such as IEXPAC questionnaire (Instrumento de Evaluación de la eXperiencia del PAciente Crónico) or Evaluation Tool of the Chronic Patient Experience and patient satisfaction (Net Promoter Score [NPS]). | Six months after inclusion of the patient
  Comparison of both strategies at the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Yun Viladomat, MD, Principal Investigator — Hospital Universitari de Bellvitge

IPD SHARING:
Plan to Share IPD: No